CLINICAL TRIAL: NCT05963633
Title: Further Forward: Future Thinking to Improve Parent-Child Relationships
Brief Title: Future Thinking to Improve Parent-Child Relationships
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Collaborators: University of Kansas (Other); University of Maryland, College Park (Other)
Responsible Party: Principal Investigator, Alyssa Vanderziel, Principal Investigator; Associate Scientist, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NARCT: 16430-01
Record Dates: First submitted 2023-07-19; First posted 2023-07-27 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-10

CONDITIONS: Behavior, Health
Keywords: episodic future thinking; delay discounting; parent-child relations; low income; substance use treatment
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Episodic Future Thinking (EFT) (Experimental): Parents who are receiving residential substance use disorder (SUD) treatment will receive an adapted episodic future thinking focused condition. Parents will meet with peer recovery coaches (PRCs) who will administer the intervention, focused on generating future, pleasant milestones with their children. The participant will also be allowed to draw or write about the scene, to help them envision it, which they will keep to refer to if they choose. After the intervention session, PRCs will check-in with parents daily over the course of two weeks to practice episodic future thinking (EFT) intervention by asking participants to further elaborate on the milestones they identified in the intervention to prompt these episodes in vivid detail.
  Interventions: Behavioral: Episodic Future Thinking (EFT)
- Episodic Recent Thinking (ERT) (Active Comparator): Parents who are receiving residential substance use disorder (SUD) treatment will receive an adapted episodic recent thinking intervention. Parents will meet with peer recovery coaches (PRCs) who will administer the intervention. During the intervention, the participant will be asked to describe in detail two things they struggled with and two things that went well that occurred during the last few days. The participant will also be allowed to draw or write about the scene, to help them envision it, which they will keep to refer to if they choose. After the intervention session, or present-oriented thinking (in the comparison condition, by asking participants to discuss an event that happened that day PRCs will check-in with parents daily over the course of two weeks to practice episodic future thinking (EFT) intervention by asking participants to further elaborate on the milestones they identified in the intervention to prompt these episodes in vivid detail.
  Interventions: Behavioral: Episodic Recent Thinking (ERT)

INTERVENTIONS:
Behavioral: Episodic Future Thinking (EFT) — The adapted episodic future thinking (EFT) intervention will focus on generation of vivid, substance-free, rewarding events that could happen in the future with their children.
  Arms: Episodic Future Thinking (EFT)
Behavioral: Episodic Recent Thinking (ERT) — In the episodic recent thinking (ERT) condition, the participant will instead describe in vivid details events that have occurred in the recent past.
  Arms: Episodic Recent Thinking (ERT)

SUMMARY:
Parents with substance use disorders are disproportionately more likely to engage in harsh physical discipline, which can lead to serious clinical outcomes, including child maltreatment and the intergenerational transmission of addictive disorders. One mechanism linking substance use and maladaptive parenting strategies is parental delay discounting, or the tendency to value smaller, immediate rewards (such as stopping children's misbehavior via physical punishment) relative to larger, but delayed rewards (like shaping adaptive child behaviors over time). This study will examine the effectiveness of a brief, episodic future thinking (EFT) intervention in a substance use treatment setting to increase parents' focus on positive, future events associated with enhancing the parent-child relationship. This study will inform broader public health efforts aimed at reducing child maltreatment and interrupting intergenerational cycles of substance abuse in traditionally underserved communities.

DETAILED DESCRIPTION:
Parents with substance use disorders (SUD) are significantly more likely to engage in harsh parenting practices, including spanking, hitting, and belittling their children, than parents without SUD. Punitive physical and emotional discipline is, in turn, associated with increased rates of child maltreatment and the subsequent intergenerational transmission of substance use disorders. Parents in residential substance use treatment facilities are among those at highest risk for perpetrating harsh and abusive parenting; yet most behaviorally based parenting interventions available within inpatient settings do not take into account the unique mechanisms linking parental substance use to harsh parenting. Specifically, parents with SUD may be at heightened risk for engaging in maladaptive parenting approaches given a tendency to prioritize immediate rewards (such as stopping a child's misbehavior using physical punishment) relative to larger, but delayed rewards (including shaping positive child behavior over a longer term). This behavioral tendency is known as delay discounting and recent findings suggest that rates of delay discounting predict parents' use of harsh physical discipline. Existing research also indicates a strong link between steeper (more problematic) rates of delay discounting and the severity of alcohol and illicit drug use across the lifespan. Thus, delay discounting may represent a specific vulnerability underlying both harsh parenting and disordered substance use. Rather than trying to decrease negative parenting practices, the focus of this study is to promote positive parent-child relationships by envisioning future-directed events. To date, no research has examined EFT in relation to parenting behaviors. Moreover, the intervention requires limited time and financial resources to implement, suggesting it may be effectively delivered in a disadvantaged community. The aims of the current study are to conduct a Stage 1 RCT (n = 72) examining the effectiveness of a brief, episodic future thinking (EFT) intervention in a substance use treatment setting serving low-income parents and additional implementation data. Participants will be randomized to receive either Episodic Future Thinking (EFT) or Episodic Recent Thinking (ERT) intervention arms. Outcomes will evaluate the effect EFT on reducing maternal delay discounting and harsh parenting and improving child clinical outcomes. Results from this case series will inform a revision of the intervention with respect to dosage and feasibility outcomes. The intervention will be delivered by peer recovery coaches who are already employed in the center.

ELIGIBILITY:
Inclusion Criteria:

1. Be the parent of a child between the ages of 6-10
2. Willing to participate in the study
3. Able to participate in written assessments and an intervention conducted in English
4. Are receiving services at Flint or Saginaw Odyssey House ("Odyssey House")
5. Be willing to receive check-ins regarding intervention content over the two weeks following the intervention
6. Can legally consent for the child to take part in the study and have regular contact with their child

Exclusion Criteria:

1. Self-disclosed active suicidality/homicidality
2. Self-disclosed current bipolar disorder, schizophrenia, or psychosis
3. Study enrollment with more than 1 child

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Delay Discounting 5 Trial Adjusted Measure | Baseline, Week 2, Week 4, Week 14
  The computer based adjusting amount discounting task uses an adjusting algorithm to determine the amount of immediately available money that is equivalent to a large sum that is delayed by seven discrete durations of time presented in a randomized order (i.e., 1 day, 1 week, 1 month, 6 months, 1 year, 5 years, and 25 years).At each delay, a choice is first presented between the delayed larger sum and a smaller sum available immediately. For each trial, the position of the delayed and immediate amounts are randomly assigned the left or right portion of the screen, and the participant chooses the preferred option by pressing the corresponding left or right response button.
Change in Consideration of Future Consequences Scale | Baseline, Week 4, Week 14
  The Consideration of Future Consequences Scale1 (CFCS-14) is a 14-item self-report questionnaire that assesses active consideration of longer-term implications of an individual's actions. Lower scores on the CFCS-14 are associated with a greater focus on immediate needs and have been found to be associated with less engagement in health behaviors1819 and greater substance use. The measure has been used extensively among adult samples and demonstrates strong reliability and validity. Research suggests modest but significant correlations with the MCQ.

SECONDARY OUTCOMES:
Change in Alabama Parenting Questionnaire Scores | Baseline, Week 4
  The Alabama Parenting Questionnaire (APQ) is a 42-item self-report measure of parenting behaviors. The questionnaire includes five subscales: (1) positive involvement with children, (2) supervision and monitoring, (3) use of positive discipline techniques, (4) consistent use of discipline, and (5) use of corporal punishment. The measure is widely used and has demonstrated excellent internal consistency and validity.

CONTACTS AND LOCATIONS:
Locations (1):
- Odyssey Village, Flint, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dassen FC, Houben K, Jansen A. Time orientation and eating behavior: Unhealthy eaters consider immediate consequences, while healthy eaters focus on future health. Appetite. 2015 Aug;91:13-9. doi: 10.1016/j.appet.2015.03.020. Epub 2015 Mar 23. PMID 25814191
- [Background] Felton JW, Kofler MJ, Lopez CM, Saunders BE, Kilpatrick DG. The emergence of co-occurring adolescent polysubstance use and depressive symptoms: A latent growth modeling approach. Dev Psychopathol. 2015 Nov;27(4 Pt 1):1367-83. doi: 10.1017/S0954579414001473. PMID 26439081
- [Background] Felton JW, Collado A, Cinader M, Lejuez CW, Chronis-Tuscano A, Yi R. Exposure to maternal depressive symptoms and growth in adolescent substance use: The mediating role of delay discounting. Dev Psychopathol. 2021 Oct;33(4):1279-1289. doi: 10.1017/S0954579420000486. PMID 32519638
- [Background] Felton JW, Collado A, Ingram KM, Doran K, Yi R. Improvement of Working Memory is a Mechanism for Reductions in Delay Discounting Among Mid-Age Individuals in an Urban Medically Underserved Area. Ann Behav Med. 2019 Oct 7;53(11):988-998. doi: 10.1093/abm/kaz010. PMID 30955043
- [Background] Lin H, Epstein LH. Living in the moment: effects of time perspective and emotional valence of episodic thinking on delay discounting. Behav Neurosci. 2014 Feb;128(1):12-9. doi: 10.1037/a0035705. PMID 24512061
- [Background] Moreland, A.M., Felton, J.F., Hanson, R.F., Jackson, C., & Dumas, J.E. (2016). The relation between parenting stress and parenting locus of control: Mechanisms of change in parenting interventions. Journal of Child and Family Studies, 25, 2046-2054.
- [Background] Stein JS, Wilson AG, Koffarnus MN, Daniel TO, Epstein LH, Bickel WK. Unstuck in time: episodic future thinking reduces delay discounting and cigarette smoking. Psychopharmacology (Berl). 2016 Oct;233(21-22):3771-3778. doi: 10.1007/s00213-016-4410-y. Epub 2016 Aug 23. PMID 27553824